CLINICAL TRIAL: NCT03667755
Title: Fast Track Recovery Feeding With a Whey Protein Infused Carbohydrate Loading Drink and Early Oral Feeding Among Surgical Gynecologic Oncology Patients: A Pragmatic Opened Labelled Trial
Brief Title: Fast Track Recovery Surgery Among Gynecologic Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, HO CHIOU YI, Dietitian, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-17-1070-36021
Record Dates: First submitted 2018-08-25; First posted 2018-09-12 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Fast Track Recovery Surgery
Keywords: pre-operation whey protein infused carbohydrate loading; early oral feeding post-operation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fast track recovery (Experimental): Participants will attend dietitian clinic to have anthropometry & dietary assessment on the same day of admission (before admission). Subjects are given a specific drink to their group on the evening prior to surgery and three hours before operation. The CHO-P group received 474ml (evening drink) or 237ml (3 hours prior to operation drink) of a lactose-free clear tea-colour fruit flavoured fluid contains 14% whey protein, 86% carbohydrates and 0% lipids. Participants fast for solids for 6 hours from the operation. Participants will be given clear fluid (2 packs Resource peach) within 24 hours post-surgery (without present of bowel sound) and reviewed by dietitian. Staff nurse in-charged will monitor anesthetic risk of drinking whey protein and ensure subject to finish specific drinks prior surgery. When they tolerated at least 500ml of clear fluids, they were given a regular solid diet.
  Interventions: Procedure: fast track recovery surgery with whey protein infused carbohydrate loading and early oral feeding
- conventional (No Intervention): Participants will attend dietitian clinic to have anthropometry & dietary assessment on the same day of admission (before admission). Participants followed conventional operation procedure whereby fasting start 12am until operation. On the first day of post-operation day, participants will be reviewed by gynaecologist and dietitian. They are allowed for clear fluid once there is bowel sound. After tolerated clear fluid, they will proceed for nourishing fluid, then soft diet and they were given a regular solid diet.

INTERVENTIONS:
Procedure: fast track recovery surgery with whey protein infused carbohydrate loading and early oral feeding — participants will be carbohydrate loaded with whey protein infused carbohydrate drink and started on early oral feeding post-operation
  Arms: fast track recovery

SUMMARY:
opened labelled randomised trial. Participants will be randomly divided into control & intervention group during admission to hospital using random numbers. Participants were randomized into two groups: the carbohydrate-protein (CHO-P) group and control (CO) group. Participants were given a specific drink to their group on the evening prior to surgery and three hours before operation. The CHO-P group received 474ml (evening drink) or 237ml (3hours prior to operation drink) of a solution contain 14% whey protein, 86% carbohydrates and 0% lipids and the CO group nil-by-mouth at 12 midnight day of operation. All participants fasted for solids for 6 hours from the operation.

DETAILED DESCRIPTION:
Candidates will attend Multidisciplinary Clinic (MDC) as appointment date for examination then they will get surgery appointment (admit to ward) 7-14 days after MDC date. Eligible patients will be identified from name list available in the electronic medical record. Selection of patient will be done by assigned research team member then she will approach and inform with study procedures to all potential candidates (selected based on inclusion and exclusion criteria) while they attend MDC during study period. Participants will be randomized into two groups: the carbohydrate-protein (CHO-P) group and conventional (CO) group during admission to hospital via random numbers which are issued by computer program. For the concepts of the CONSORT flow diagram are followed [50]. The Patient Information Consent Form will be given to identify eligible subjects who agreed to be recruited in the study. Subjects are allowed to bring back consent form if she keen to seek advice from family member.

Carbohydrate-protein group: Participants will attend dietitian clinic to have anthropometry & dietary assessment on the same day of admission (before admission). Subjects are given a specific drink to their group on the evening prior to surgery and three hours before operation. The CHO-P group received 474ml (evening drink) or 237ml (3 hours prior to operation drink) of a lactose-free clear tea-colour fruit flavoured fluid contains 14% whey protein, 86% carbohydrates and 0% lipids. Participants fast for solids for 6 hours from the operation. Participants will be given clear fluid (2 packs Resource peach) within 24 hours post-surgery (without present of bowel sound) and reviewed by dietitian. Staff nurse in-charged will monitor anesthetic risk of drinking whey protein and ensure subject to finish specific drinks prior surgery. When they tolerated at least 500ml of clear fluids, they were given a regular solid diet.

Conventional group: Participants will attend dietitian clinic to have anthropometry & dietary assessment on the same day of admission (before admission). Participants followed conventional operation procedure whereby fasting start 12am until operation. On the first day of post-operation day, participants will be reviewed by gynaecologist and dietitian. They are allowed for clear fluid once there is bowel sound. After tolerated clear fluid, they will proceed for nourishing fluid, then soft diet and they were given a regular solid diet.

On the day of operation and on the first day of post-operative day, blood samples are collected for hemoglobin, renal profile, albumin and C-reactive protein. Biochemical data will be record from electronic medical record. Upon discharge, all participants will be sent to dietitian clinic to assess anthropometry and dietary data.

ELIGIBILITY:
Inclusion Criteria:

* who diagnosed with Gynecologic Cancer stage 1 to stage 4
* candidates for elective operation treatments
* Malaysian aged more than 18 years old

Exclusion Criteria:

* Not a candidate for elective operation treatments
* Aged <18 years old
* Diagnosed with Diabetes Mellitus/Chronic Kidney Disease/Heart disease/Chronic liver disease
* Allergy to milk/soy/whey protein
* participate other intervention study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
length of post-operative hospital stay | throughout hospitalization (up to 2 weeks)
  period of hospitalization after operation to discharged
length of clear fluid toleration | throughout hospitalization (up to 1 week)
  period of clear fluid toleration post-operation
length of solid food toleration | throughout hospitalization (up to 2 weeks)
  period of solid food toleration post-operation

SECONDARY OUTCOMES:
height | throughout hospitalization (up to 2 weeks)
  outcomes will be measured once (admission). Measurement in meter.
dietary intake trend during hospitalization | daily energy and protein intake throughout hospitalization (up to 2 weeks)
  kilocalories for energy; gram for protein
inflammatory effect | on day of operation (before operation and 12 hours after operation)
  C-reactive protein in mg/L
post-operative complications | throughout hospitalization (up to 2 weeks)
  infection (yes/no), ileus (yes/no), nausea (yes/no), vomiting (yes/no)
re-admission | 1 month post-operation
  re-admission within 1 month post operation
muscle mass | throughout hospitalization (up to 2 weeks)
  Assessment will be measured twice (upon admission and upon discharged). Unit of measure for muscle mass is in kilogram
weight | throughout hospitalization (up to 2 weeks)
  outcomes will be measured twice (admission and upon discharged). Units of Measure such as weight in kilogram
Body Mass Index | throughout hospitalization (up to 2 weeks)
  outcomes will be measured twice (admission and upon discharge). Units of Measure BMI in kg/m^2
handgrip strength | throughout hospitalization (up to 2 weeks)
  outcomes will be measured twice (admission and upon discharged). Units of Measure is handgrip strength in kilogram

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Putrajaya, Putrajaya, Malaysia

REFERENCES:
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396
- [Derived] Ho CY, Ibrahim Z, Abu Zaid Z, Mat Daud Z', Md Yusop NB. Fast-track- recovery surgery with a whey-protein-infused carbohydrate-loading drink pre-operatively and early oral feeding post-operatively among surgical gynaecological cancer patients: study protocol of an open-labelled, randomised controlled trial. Trials. 2020 Jun 16;21(1):533. doi: 10.1186/s13063-020-04462-4. PMID 32546217

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03667755/Prot_SAP_ICF_000.pdf